CLINICAL TRIAL: NCT00641212
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Study of the Effect of Long-Term Treatment With Rhinocort Aqua (Budesonide) Nasal Spray in Children With Perennial Allergic Rhinitis.
Brief Title: Children, Perennial Allergic Rhinitis (PAR), l-t Growth
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SD-005-0414; D5360C00414
Record Dates: First submitted 2008-03-18; First posted 2008-03-24 (Estimated); Last update posted 2009-03-25 (Estimated); Status verified 2009-03

CONDITIONS: Perennial Allergic Rhinitis
Keywords: Allergic rhinitis; Perennial allergic rhinitis; Paediatric; Growth; budesonide; Rhinocort AQUA
MeSH Terms: conditions — Rhinitis, Allergic, Perennial; Rhinitis, Allergic | interventions — Budesonide

ARMS (2):
- 1 (Experimental): Budesonide
  Interventions: Drug: Budesonide
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Budesonide
  Other Names: Rhinocort AQUA
  Arms: 1
Drug: Placebo
  Arms: 2

SUMMARY:
The purpose of this study is to compare the effect of Rhinocort nasal spray with placebo on growth in children with perennial allergic rhinitis over 12 months.

ELIGIBILITY:
Inclusion Criteria:

* In the opinion of the investigator, is a candidate for treatment with nasal steroids based on a history of either a) inadequate control of symptoms with antihistamines, decongestants and/or immunotherapy, or b) prior successful treatment with nasal steroids.
* A documented history of at least one year of perennial allergic rhinitis.
* A positive response to a skin prick test for perennial allergens that must be present in the subject's environment.
* Height and weight within normal limits.

Exclusion Criteria:

* Any disease which may affect growth
* Sexual development later than Tanner stage I.
* Nasal candidiasis, rhinitis medicamentosa, acute or chronic sinusitis, influenza, upper respiratory tract infection or structural abnormalities of the nose (e.g., septal deviation, nasal polyps) symptomatic enough to cause significant nasal obstruction as judged by the investigator.

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 209 (Estimated)
Dates: Start 2000-01; Primary Completion 2003-04 (Actual); Study Completion 2003-04 (Actual)

PRIMARY OUTCOMES:
Change in height over a 12 month period | 3 monthly

SECONDARY OUTCOMES:
Change in growth velocity over a 12 month period. | 3 monthly
Other safety - assessed by adverse event query | 3 monthly

CONTACTS AND LOCATIONS:
Overall Officials: Bertil Andersson, Study Director — AstraZeneca